CLINICAL TRIAL: NCT02523209
Title: Analysis of Bone Microarchitecture With HR-pQCT of Patients With Chronic Kidney Disease (CKD) Candidates for Renal Transplantation - A Monocentric Study
Brief Title: Analysis of Bone Microarchitecture With HR-pQCT of Patients With Chronic Kidney Disease (CKD) Candidates for Renal Transplantation
Acronym: TRANSBONE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1408080
Record Dates: First submitted 2015-07-15; First posted 2015-08-14 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Chronic Kidney Diseases; Hyperparathyroidism, Secondary
Keywords: Osteoporosis; chronic kidney disease; kidney transplantation; fracture risk
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bone quality and quantity: measure of bone quality and quantity parameters by HRpQCT and by DEXA
  Interventions: Device: HR-pQCT; Device: DEXA

INTERVENTIONS:
Device: HR-pQCT — HR-pQCT (High Resolution peripheral micro Computerized Tomography) is a device used for 3D bone measurements at the tibia and the radius levels in humans.
Device: DEXA — The Lunar DEXA (Dual Energy X-ray Absorptiometry) is a third generation multi-captor DEXA (Dual Energy X-ray Absorptiometry) device that allows short duration measurements ( <15 min). It measures Bone Mineral Density at the spine (L1-L4) and the femoral neck

SUMMARY:
While the duration of renal transplant function has increased over the last decade kidney transplanted patients (KTP) still exhibit a fracture risk 4 times higher than in the general population. Fracture risk remains increased despite the improvement of immunosuppressive therapies (IST) that allowed the reduction of steroid administration. Potential explanations for this could be 1) that Chronic Kidney Disease (CKD) induces renal osteodystrophy that occurs before kidney transplanted, impairs bone metabolism and promotes bone fragility ; 2) that kidney transplanted patients are older and older (14% of kidney transplanted patients were older than 70 in 2011 in France), ageing being a major risk factor for fractures 3) IST, besides steroid, may have deleterious effects on bone and 4) that secondary hyperparathyroidism, a risk factor of fractures, persists after kidney transplanted . Thus, the pathophysiology and epidemiology of bone fragility of kidney transplanted patient remains insufficiently characterized. Despite these data, and contrarily to what is done for patients candidates for cardiac transplantation, there is no general consensus for performing bone evaluation before kidney transplanted . Thus it's necessary to individualize the management of bone fragility and prevent fractures according to strategies that remain to be defined, provided that patients at risk are better detected.

DETAILED DESCRIPTION:
Bone fragility is determined by quantitative parameters (bone mass) and qualitative parameters including macro- and micro-architecture (especially cortical porosity and thickness). The Dual Energy X-ray Absorptiometry (DEXA ) measurement of Bone Mineral Density (BMD) is a robust predictor of fracture risk in the non-uremic population. Micro and macro-architecture can be measured with High Resolution peripheral micro Computerized Tomography (HRpQCT) at the ankle and the wrist . Some recent studies suggested that HRpQCT could be a better fracture predictor than DEXA in uremic populations. In this context, the aim of our project is to describe in a cross sectional study the bone status of CKD patients, candidates for kidney transplanted . It will be 1) calculated the prevalence of cortical osteoporosis as assessed by cortical thickness at the ankle and the wrist (primary end point), 2) analyzed other HRpQCT microarchitecture quantitative parameters and 3) defined the biological and clinical factors associated with bone degradation (secondary endpoints). This population will be compared to age and sex matched normal subjects (collaboration with Pr Rizzoli, Geneva, Switzerland). The DEXA and HRpQCT will be compared for detection of patients at risk for fracture.

ELIGIBILITY:
Inclusion Criteria:

* Serum parathyroidal Hormon (PTH ) > 65pg/ml
* Stage 5 or 5D Chronic Kidney Disease patients
* Patient registered (or on the verge of being registered) on the KT waiting list at St-Etienne Hospital, France
* Written consent of patient

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with end stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with cortical osteoporosis | Day1
  A Cortical osteoporosis is a composite outcome measured with two devices : HR-pQCT and DEXA parameters measured with HR-pQCT on ankle (tibia) and wrist (radius) are : Cortical thickness (mm). Parameters measured with DEXA on spine and femoral neck are : Bone Mineral Density (BMD, g/cm2)

SECONDARY OUTCOMES:
clinical and biological factors associated with bone degradation | day 1
  clinical and biological factors are a composite outcome : Clinical parameters measured are : dialysis vintage, age, transplantation history , sex, Immunosuppressive Therapies, steroid dose, parathyroidectomy history, Biological parameters measured are Calcium, Phosphorus, Parathormone, bicarbonates, albumin, Bone alkaline phosphatase.
  Bone degradation is a composite measure : parameters measured with HR-pQCT on ankle (tibia) and wrist (radius) are :
  Cortical thickness (mm), Total mineral volumetric density (mg/ccm HA), trabecular mineral volumetric density (mg/ccm HA), Cortical mineral volumetric density (mg/ccm HA), Trabecular Number (1/mm), Trabecular thickness (mm), Trabecular Separation (mm), Mean distance between trabecular (mm) Parameters measured with DEXA on spine and femoral neck are : Bone Mineral Density (BMD, g/cm2), T-Score, Z-Score, Trabecular bone score (TBS).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène LAFAGE-PROUST, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France